CLINICAL TRIAL: NCT04490629
Title: A Prospective, Multi-center, Randomized, Parallel-controlled Clinical Trial Evaluating the Efficacy and Safety of Lyoplant Onlay in Repairing Cerebral Dura Mater
Brief Title: The Efficacy and Safety of a Latest Dural Substitute
Acronym: ESLO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-126
Record Dates: First submitted 2020-07-16; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Cerebrospinal Fluid Leak
Keywords: Dura Mater; Cerebrospinal Fluid Leak
MeSH Terms: conditions — Cerebrospinal Fluid Leak

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DURAFORM (Other): DURAFORM was used in repairing cerebral dura mater.
  Interventions: Device: DURAFORM
- Lyoplant Onlay (Experimental): Lyoplant Onlay was used in repairing cerebral dura mater.
  Interventions: Device: Lyoplant Onlay

INTERVENTIONS:
Device: Lyoplant Onlay — Lyoplant Onlay is a kind of latest artificial Dura Mater
  Arms: Lyoplant Onlay
Device: DURAFORM — DURAFORM is a kind of conventional artificial Dura Mater
  Arms: DURAFORM

SUMMARY:
This prospective, multi-center, randomized, parallel-controlled clinical trial was designed to evaluate the efficacy and safety of Lyoplant Onlay in repairing cerebral dura mater. DURAFORM was regarded as the control group. a total of 80 patients were randomized into experimental and control group (1:1).Data were collected on complications resulting in CSF leaks, surgical site infections, instrument performance parameterized other neurological complications within 30 days. Surgeons also provided data on the ease of use of the dural sealing techniques, as well as preparation and application times. The above-mentioned date were used to evaluate the efficacy and safety of Lyoplant Onlay .

ELIGIBILITY:
Inclusion Criteria:

* Any patient between the ages of 18 and 75 years scheduled for elective cranial surgery involving a dural incision.
* Dural defects and surgical incision was classifed as level 1

Exclusion Criteria:

* local or systemic infection.
* patients with known allergy to Equipment components
* a history of traumatic head injury
* a compromised immune system or autoimmune disease
* patients who should not participate based on the surgeon's opinion
* patients participating in any other drug or device trial.
* expected survival time <12 months
* underwent chemoradiotherapy 3 months before randomization
* uncontrolled diabetes and malignant tumor
* women who were pregnant, lactating, or wished to become pregnant during the study;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
surgical successful rate | at 30 days post surgery
  proportion of treated patients free of CSF leak diagnosed by physical examination, biochemical assay, or imaging study within 30 d of the surgical procedure.

SECONDARY OUTCOMES:
neurosurgical complication | 2 days post surgery/10 days post surgery/at 30 days post surgery
  Incidence of intracranial infection at 2 days after operation，at discharge，and at 30 days after operation

CONTACTS AND LOCATIONS:
Overall Officials: jianmin zhang, M.D., Principal Investigator — Department of neurosurgery
Locations (1):
- Jianmin Zhang, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
The committee will debate whether to share IPD depending on the circumstances. Because some patients are unwilling to make their condition known.